CLINICAL TRIAL: NCT04488692
Title: The Effect of Two Models of an Early Intervention Program on Functional Recovery at Three Months to Acute Stroke Patients: A Randomized Controlled Trial
Brief Title: Early Functional Training in Acute Stroke Inpatient Ward
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chung Shan Medical University (Other)
Responsible Party: Principal Investigator, Ching-Yi Wang, Professor, Chung Shan Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CS19166
Record Dates: First submitted 2020-07-21; First posted 2020-07-28 (Actual); Last update posted 2022-10-25 (Actual); Status verified 2022-10

CONDITIONS: Acute Stroke
MeSH Terms: conditions — Stroke | interventions — Early Intervention, Educational

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Model 1 (Experimental): Participants will receive 2 sessions of functional training per day, 15-min per session.
  Interventions: Other: Early intervention (Mobility functional training)
- Model 2 (Active Comparator): Participants will receive 1 session of functional training and 1 session of sham intervention (therapist visiting and education) per day, 15-min per session.
  Interventions: Other: Early intervention (Mobility functional training); Other: Sham intervention

INTERVENTIONS:
Other: Early intervention (Mobility functional training) — functional training focused on mobility (bed mobility, sitting balance, standing balance, and ambulation)
Other: Sham intervention — friendly visit and education
  Arms: Model 2

SUMMARY:
To investigate the difference between two models of an early intervention program (focused on mobility function) in the functional recovery 3 months post stroke in a group of patients with acute ischemic stroke while in acute inpatient ward hospitalization.

DETAILED DESCRIPTION:
Patients with acute stroke admit into an acute inpatient ward who meet study criteria and provide institutional-reviewed consent form will be randomly assigned into either model 1 or model 2 of an early functional training program. Participants in model 1 group will receive 2 sessions of functional training per day whereas those in model 2 group will receive 1 session of functional training and 1 session of friendly visit and education per day. The following outcomes will be measured at admission, at discharge and at 3 months post stroke: Barthel index (BI), Postural Assessment Scale for Stroke (PASS), Mobility Scale for Acute Stroke (MASA), and usual gait speed (UGS). The rater is blinded to participants' group membership.

ELIGIBILITY:
Inclusion Criteria:

* patient with acute ischemic stroke / ICH
* referred for early rehabilitation,
* aged 20 years or more,

Exclusion Criteria:

* able to walk independently and safely at admission,
* unable to understand three simple comments,
* unable to recovery even with appropriate medical management,
* serious condition require ICU care,
* terminal illness for hospice care,
* waiting to transfer to long term care facilities

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2022-03-04 (Actual); Study Completion 2022-03-04 (Actual)

PRIMARY OUTCOMES:
Postural Assessment Scale for Stroke Patient (PASS) | Baseline
  The total score range is 0 to 36 points. Higher score indicate better performance.
Postural Assessment Scale for Stroke Patient (PASS) | up to 2 weeks
  The total score range is 0 to 36 points. Higher score indicate better performance.
Postural Assessment Scale for Stroke Patient (PASS) | at 3 months post stroke
  The total score range is 0 to 36 points. Higher score indicate better performance.
Barthel index (BI) | Baseline
  The total score range is 0 to 100 points. Higher score indicate better performance.
Barthel index (BI) | up to 2 weeks
  The total score range is 0 to 100 points. Higher score indicate better performance.
Barthel index (BI) | at 3 months post stroke
  The total score range is 0 to 100 points. Higher score indicate better performance.

SECONDARY OUTCOMES:
Usual gait speed | Baseline
  meters per second. Higher score indicate better performance.
Usual gait speed | up to 2 weeks
  meters per second. Higher score indicate better performance.
Usual gait speed | at 3 months post stroke
  meters per second. Higher score indicate better performance.
Mobility Scale for Acute Stroke (MSAS) | Baseline
  The total score range is 6 to 36 points. Higher score indicate better performance.
Mobility Scale for Acute Stroke (MSAS) | up to 2 weeks
  The total score range is 6 to 36 points. Higher score indicate better performance.
Mobility Scale for Acute Stroke (MSAS) | at 3 months post stroke
  The total score range is 6 to 36 points. Higher score indicate better performance.

CONTACTS AND LOCATIONS:
Overall Officials: Ching-Yi Wang, PhD, Principal Investigator — Chung Shan Medical University
Locations (1):
- Chung Shan Medical University Hospital, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Adams HP Jr, Brott TG, Crowell RM, Furlan AJ, Gomez CR, Grotta J, Helgason CM, Marler JR, Woolson RF, Zivin JA, et al. Guidelines for the management of patients with acute ischemic stroke. A statement for healthcare professionals from a special writing group of the Stroke Council, American Heart Association. Circulation. 1994 Sep;90(3):1588-601. doi: 10.1161/01.cir.90.3.1588. No abstract available. PMID 8087974
- [Background] Bernhardt J, Churilov L, Ellery F, Collier J, Chamberlain J, Langhorne P, Lindley RI, Moodie M, Dewey H, Thrift AG, Donnan G; AVERT Collaboration Group. Prespecified dose-response analysis for A Very Early Rehabilitation Trial (AVERT). Neurology. 2016 Jun 7;86(23):2138-45. doi: 10.1212/WNL.0000000000002459. Epub 2016 Feb 17. PMID 26888985
- [Background] Bernhardt J, Dewey H, Thrift A, Collier J, Donnan G. A very early rehabilitation trial for stroke (AVERT): phase II safety and feasibility. Stroke. 2008 Feb;39(2):390-6. doi: 10.1161/STROKEAHA.107.492363. Epub 2008 Jan 3. PMID 18174489
- [Background] Diserens K, Moreira T, Hirt L, Faouzi M, Grujic J, Bieler G, Vuadens P, Michel P. Early mobilization out of bed after ischaemic stroke reduces severe complications but not cerebral blood flow: a randomized controlled pilot trial. Clin Rehabil. 2012 May;26(5):451-9. doi: 10.1177/0269215511425541. Epub 2011 Dec 2. PMID 22144725
- [Background] Indredavik B, Bakke F, Solberg R, Rokseth R, Haaheim LL, Holme I. Benefit of a stroke unit: a randomized controlled trial. Stroke. 1991 Aug;22(8):1026-31. doi: 10.1161/01.str.22.8.1026. PMID 1866749
- [Background] Krakauer JW, Carmichael ST, Corbett D, Wittenberg GF. Getting neurorehabilitation right: what can be learned from animal models? Neurorehabil Neural Repair. 2012 Oct;26(8):923-31. doi: 10.1177/1545968312440745. Epub 2012 Mar 30. PMID 22466792
- [Background] Kwakkel G, van Peppen R, Wagenaar RC, Wood Dauphinee S, Richards C, Ashburn A, Miller K, Lincoln N, Partridge C, Wellwood I, Langhorne P. Effects of augmented exercise therapy time after stroke: a meta-analysis. Stroke. 2004 Nov;35(11):2529-39. doi: 10.1161/01.STR.0000143153.76460.7d. Epub 2004 Oct 7. PMID 15472114
- [Background] Langhorne P, Collier JM, Bate PJ, Thuy MN, Bernhardt J. Very early versus delayed mobilisation after stroke. Cochrane Database Syst Rev. 2018 Oct 16;10(10):CD006187. doi: 10.1002/14651858.CD006187.pub3. PMID 30321906
- [Background] Langhorne P, Wu O, Rodgers H, Ashburn A, Bernhardt J. A Very Early Rehabilitation Trial after stroke (AVERT): a Phase III, multicentre, randomised controlled trial. Health Technol Assess. 2017 Sep;21(54):1-120. doi: 10.3310/hta21540. PMID 28967376
- [Background] Langhorne P, Stott D, Knight A, Bernhardt J, Barer D, Watkins C. Very early rehabilitation or intensive telemetry after stroke: a pilot randomised trial. Cerebrovasc Dis. 2010;29(4):352-60. doi: 10.1159/000278931. Epub 2010 Jan 30. PMID 20130401
- [Background] Lee KB, Lim SH, Kim KH, Kim KJ, Kim YR, Chang WN, Yeom JW, Kim YD, Hwang BY. Six-month functional recovery of stroke patients: a multi-time-point study. Int J Rehabil Res. 2015 Jun;38(2):173-80. doi: 10.1097/MRR.0000000000000108. PMID 25603539
- [Background] Stinear CM, Byblow WD, Ackerley SJ, Smith MC, Borges VM, Barber PA. Proportional Motor Recovery After Stroke: Implications for Trial Design. Stroke. 2017 Mar;48(3):795-798. doi: 10.1161/STROKEAHA.116.016020. Epub 2017 Jan 31. PMID 28143920
- [Background] Sundseth A, Thommessen B, Ronning OM. Early mobilization after acute stroke. J Stroke Cerebrovasc Dis. 2014 Mar;23(3):496-9. doi: 10.1016/j.jstrokecerebrovasdis.2013.04.012. Epub 2013 May 13. PMID 23680682
- [Background] Verheyden G, Nieuwboer A, De Wit L, Thijs V, Dobbelaere J, Devos H, Severijns D, Vanbeveren S, De Weerdt W. Time course of trunk, arm, leg, and functional recovery after ischemic stroke. Neurorehabil Neural Repair. 2008 Mar-Apr;22(2):173-9. doi: 10.1177/1545968307305456. Epub 2007 Sep 17. PMID 17876069
- [Background] Wade DT, Wood VA, Hewer RL. Use of hospital resources by acute stroke patients. J R Coll Physicians Lond. 1985 Jan;19(1):48-52. No abstract available. PMID 3973842
- [Background] Xu T, Yu X, Ou S, Liu X, Yuan J, Chen Y. Efficacy and Safety of Very Early Mobilization in Patients with Acute Stroke: A Systematic Review and Meta-analysis. Sci Rep. 2017 Jul 26;7(1):6550. doi: 10.1038/s41598-017-06871-z. PMID 28747763